CLINICAL TRIAL: NCT06688877
Title: Einfluss Der Kombination Von Musik Und Noise Cancelling Als nichtmedikamentöse Unterstützung Bei Angst Und Unwohlsein während Der Weisheitszahnentfernung
Brief Title: The Study is About the inﬂuence of the Combination of Music and Noise Cancelling as a Non-pharmacological Aid in Reducing Anxiety and Discomfort During Wisdom Tooth Removal. The Level of Fear is Measured by a Questionnaire Which the Patients Answer Twice and a Measurement of the Heartbeat
Status: Not yet recruiting | Type: Observational
Sponsor: Sigmund Freud PrivatUniversitat (Other)
Responsible Party: Sponsor
Other Study IDs: 834-2023
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Fear Anxiety; Wisdom Tooth Removal; Heart Rate
Keywords: fear level; wisdom teeth removal; noise reduction by music and noise cancelling
MeSH Terms: interventions — Heart Rate; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Controlgroup: No headphones, no music, no noise cancelling (no additional treatment): Experimental group 1: headphones with activated noise cancelling
  Interventions: Device: heart rate measurement; Other: Questionnaire
- Experimental group 2: headphones with activated noise cancelling and soft 60 bpm music
  Interventions: Device: headphones with activated noise cancelling and soft 60 bpm musc; Device: heart rate measurement; Other: Questionnaire
- Experimental group 1: headphones with activated noise cancelling
  Interventions: Device: headphones with activated noise cancelling; Device: heart rate measurement; Other: Questionnaire

INTERVENTIONS:
Device: headphones with activated noise cancelling — noise cancelling is new
  Groups: Experimental group 1: headphones with activated noise cancelling
Device: headphones with activated noise cancelling and soft 60 bpm musc — noise cancelling is new
  Groups: Experimental group 2: headphones with activated noise cancelling and soft 60 bpm music
Device: heart rate measurement — three times (before, during and after surgery)
Other: Questionnaire — two times (before and after surgery)

SUMMARY:
The goal of this clinical trial is to learn if the reduction of the noises (through head phones with music and noise cancelling) that occur during wisdom teeth removal, leads to a significant reduction in fear levels in patients compared to patients who do not have any noise reduction. The main questions it aims to answer are:

Do music and noise cancelling help patients to have less fear during wisdom teeth removal surgery by reducing the sounds of the surgery? Is there a difference between just the noise cancelling function or is it better to combine noise cancelling and music together?

Participants will:

Just come to their regular appointment (wisdom teeth removal) to our clinic, no follow ups needed. All participants will answer one questionnaire before and one after the surgery. All of them will have their rate of heartbeat measured for three times (before, during and after surgery, measured by a puls oximeter on the finger). They will be allocated to one of the three study groups (no headphones, headphones with noise cancelling or headphones with noise cancelling and music).

DETAILED DESCRIPTION:
The headphones that will be used are Sennheiser Overear Headphones with modern noise cancelling function.

Pulse Oximeter is by BRAUN and CE-certified.

Observational Study Model: Randomised controlled, unblinded clinical trial, parallel group design

Sampling method: randomisation by a online randomizer tool

ELIGIBILITY:
Inclusion Criteria:

* willing to participate in the clinical trial, understood and signed the information sheet

Exclusion Criteria:

* younger than 18 years old
* hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have to get their wisdom tooth removed at the dental clinic of the Sigmund Freud Private University of Vienna, aged minimum 18 years old, no hearing impairment, want to take part in the clinical trial.
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2025-06-29 (Estimated); Study Completion 2025-06-29 (Estimated)

PRIMARY OUTCOMES:
Result of the questionnaire | Answering the first questionnaire to answering the second questionnaire happens both on the same day, right before and right after the surgery.
  The primary outcome measure is the result of the questionnaire, which the probands answer two times, before and after the surgery. The score of these two will be summarized for a final result of each patient.

SECONDARY OUTCOMES:
Measurement of the heart rate | All three measurements happen on the same day. Before, during and after the surgery, no follow up.
  The Secondary Outcome Measure is the Measurement of the heart rate. This will happen three times: right before, right after and at a set point during the surgery. The pulse oximeter is clipped on a finger of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Zahnklinik der SFU Wien / Dental clinic of the Sigmund Freud private univeristy Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No